CLINICAL TRIAL: NCT02330991
Title: A Trial of One-week on/One-week Off Temozolomide Versus Continuous Dose-Intense Temozolomide in Patients With Glioblastoma Multiforme at First Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Junping Zhang, Chief Physician, Beijing Sanbo Brain Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014062501
Record Dates: First submitted 2014-12-30; First posted 2015-01-05 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Glioblastoma
Keywords: glioblastoma; relapse; Temozolomide; glioblastoma at first relapse
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Temozolomide

ARMS (2):
- Arm1 ,one-week on/one-week off regimen (Experimental): One-week on/one-week off regimen is administered for 12 cycles of 28 days. Arm 1 receives temozolomide 150 mg/m2 daily during days 1 to 7 and 15 to 21 of each cycle.Treatment will continue until tumor progression, development of excessive toxicity, withdrawal of consent, or completion of 12 cycles.
  Interventions: Drug: Temozolomide
- Arm 2,continuous dose-intense regimen (Experimental): Continuous dose-intense regimen is administered for 12 cycles of 28 days .Arm 2 receives temozolomide 50mg/m2 daily during days 1 to 28 of each cycle. Treatment will continue until tumor progression, development of excessive toxicity, withdrawal of consent, or completion of 12 cycles.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide
  Other Names: Temodal

SUMMARY:
The purpose of this study is to evaluate the clinical benefit and safety of two different Dose-Intense temozolomide regimens（one-week on/one-week off regimen versus continuous dose-intense regimen）in patients with glioblastoma at first relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histopathologically-confirmed, supratentorial, glioblastoma.
2. Participants must have received first-line treatment regimen consisting of RT plus concomitant temozolomide followed by adjuvant temozolomide.
3. Participants must be first recurrence or progression of glioblastoma after first-line treatment regimen.
4. Participants must have demonstration of recurrent disease on MRI following prior therapy.
5. Participants must have bi-dimensionally measurable disease with a minimum measurement of 1 cm in one dimension on MRI performed within 14 days prior to first treatment. If receiving corticosteroids, participants must be on a stable or decreasing dose of corticosteroids for at least 5 days prior to baseline MRI.
6. Participants must have developed progressive disease after receiving prior therapy and must have an interval of at least 12 weeks from the completion of radiation and concomitant temozolomide therapy to study entry (unless progressive tumor growth is outside the radiation field or there is histopathological confirmation of recurrent tumor)
7. Age 18-75 years old.
8. Life expectancy of at least 12 weeks.
9. Karnofsky performance status at least 60
10. Participants must be able to adhere to the dosing and visit schedules, and agree to record medication times, concomitant medications, and adverse events (AEs) accurately and consistently in a daily diary.
11. 20 paraffinsections of glioblastoma tissue must be available.
12. Participants must have normal organ and marrow function as defined below: leukocytes >4.0×10^9/L，platelets >100×10^9/L，Hemoglobin > 10 g/dl，Serum creatinine< 1.5-fold upper normal range，AST and ALT <2-fold upper normal range, Alkaline phosphatase < 3-fold upper normal range.
13. Female and male subjects of childbearing potential must agree to use a medically accepted method of adequate contraception.

Exclusion Criteria:

1. Treatment with any chemotherapy other than temozolomide prior to enrollment.
2. Progressive or recurrent glioblastoma documented by MRI earlier than 12 weeks after completion of radiotherapy.
3. History of any other cancer.
4. HIV infection.
5. Women who are pregnant or breast feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Progress-Free Survival at 6 months (PFS6) | 6 months

SECONDARY OUTCOMES:
Overall Survival(OS) | 2 years
Progression free survival | 2 years
Objective Response Rate | up to 52 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Junping Zhang, MD, Principal Investigator — Beijing Sanbo Brain Hospital